CLINICAL TRIAL: NCT00619697
Title: Comparison of Efficacy and Safety of Biphasic Insulin Aspart 30 Plus Metformin With Insulin Glargine Plus Glimepiride in Type 2 Diabetes
Brief Title: Efficacy and Safety of Biphasic Insulin Aspart 30 in Combination With Metformin in Type 2 Diabetes
Acronym: EUROMIX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1564
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Glargine; Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
  Other Names: BIASP; NovoMix 30; NovoLog 70/30 Mix
Drug: insulin glargine
Drug: metformin
Drug: glimepiride

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the efficacy on blood glucose control in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 6 months
* Insulin naive. Short term insulin treatment (7 days or less within the last 6 months) is allowed
* Previous treatment with oral antidiabetic drugs for at least 4 months
* Judged by the investigator to be eligible for an insulin analogue plus oral antidiabetic drug treatment regimen
* BMI below 40 kg/m2
* HbA1c between 7-12%
* Able and willing to perform self-plasma glucose monitoring

Exclusion Criteria:

* The receipt of any other investigational drug within 4 weeks before screening
* A history of drug or alcohol abuse within the last 12 months
* Severe, uncontrolled hypertension
* Known or suspected allergy to trial products or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2003-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 26 weeks of treatment

SECONDARY OUTCOMES:
HbA1c | after 16 weeks of treatment
Plasma glucose profiles
Change in body mass index
Incidence of hypoglycaemic episodes
Safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (49):
- Austria (8):
  - Novo Nordisk Investigational Site, Ebreichsdorf
  - Novo Nordisk Investigational Site, Feldkirch
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Horn
  - Novo Nordisk Investigational Site, Oberpullendorf
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Villach
  - Novo Nordisk Investigational Site, Waidhofen A.d. Thaya
- Czechia (2):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Liberec
- Germany (26):
  - Novo Nordisk Investigational Site, Augsburg
  - Novo Nordisk Investigational Site, Castrop-Rauxel
  - Novo Nordisk Investigational Site, Deggingen
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Erlangen
  - Novo Nordisk Investigational Site, Eschweiler
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Fulda
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Herne
  - Novo Nordisk Investigational Site, Kippenheim
  - Novo Nordisk Investigational Site, Lauffen am Neckar
  - Novo Nordisk Investigational Site, Leverkusen
  - Novo Nordisk Investigational Site, Ludwigsburg
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Mannheim
  - Novo Nordisk Investigational Site, Marburg
  - Novo Nordisk Investigational Site, Mülheim
  - Novo Nordisk Investigational Site, Neunkirchen
  - Novo Nordisk Investigational Site, Ostercappeln
  - Novo Nordisk Investigational Site, Pritzwalk
  - Novo Nordisk Investigational Site, Rosenheim
  - Novo Nordisk Investigational Site, Viernheim
  - Novo Nordisk Investigational Site, Weil der Stadt
  - Novo Nordisk Investigational Site, Weiskirchen
  - Novo Nordisk Investigational Site, Witten
- Hungary (3):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Eger
  - Novo Nordisk Investigational Site, Szekszárd
- Poland (5):
  - Novo Nordisk Investigational Site, Częstochowa
  - Novo Nordisk Investigational Site, Gdynia
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Otwock
  - Novo Nordisk Investigational Site, Poznan
- Slovakia (2):
  - Novo Nordisk Investigational Site, L'ubochna
  - Novo Nordisk Investigational Site, Martin
- Slovenia (3):
  - Novo Nordisk Investigational Site, Celje
  - Novo Nordisk Investigational Site, Ljubljana
  - Novo Nordisk Investigational Site, Maribor

REFERENCES:
- [Result] Kann PH, Wascher T, Zackova V, Moeller J, Medding J, Szocs A, Mokan M, Mrevlje F, Regulski M. Starting insulin therapy in type 2 diabetes: twice-daily biphasic insulin Aspart 30 plus metformin versus once-daily insulin glargine plus glimepiride. Exp Clin Endocrinol Diabetes. 2006 Oct;114(9):527-32. doi: 10.1055/s-2006-949655. PMID 17115351
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com